CLINICAL TRIAL: NCT01420315
Title: The Prevalence of Vitamin D Deficiency in Patients With Alzheimer's Disease: a Crosssectional Multicenter Study in Turkey
Brief Title: The Prevalence of Vitamin D Deficiency in Patients With Alzheimer's Disease
Acronym: DEVIT-ALZ
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Mehmet Ilkin Naharci, Assistant professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: VDGT-01; G-123456789 (Other: Gulhane Medical Training School)
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease
Keywords: vitamin D; deficiency; alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Recent studies indicate that there is a relationship between cognitive decline and vitamin D deficiency. Up to now, no study has investigated the prevalence of vitamin d deficiency in patient with Alzheimer's disease. Our aim is to investigate the prevalence of vitamin D deficiency and analysis the associated characteristics in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Vitamin D has many physiological functions via skeletal and extra-skeletal effects. Nowadays, it is well known that vitamin d deficiency causes to an increase in disease burden. As the role of vitamin D, the maintenance of balance, the improvement of muscle power, and the augmentation of innate immunity were proven. Some recent studies showed that vitamin D deficiency associates with cardiovascular diseases, autoimmune diseases, and the risk of cancer.

Vitamin D carries out your functions by vitamin d receptors (VDR) located in many cells. Brain neurons and glial cells are including VDR's. It is presumed that the functions of vitamin d in neurons are the regulation of neurotransmission, neuron protection, and immunomodulation. Also,vitamin D has a role in brain development and maturation. Except the functions in central nerve system, vitamin D has effects on peripheral nerve system. It was reported that nerve transduction velocity decreased in vitamin d deficiency.

Vitamin D deficiency and Alzheimer's disease are major public health problems that their incidences increase in advanced ages.Recent studies indicate that there is a relationship between cognitive decline and vitamin D deficiency. VDR receptors in brain specially in hippocampus, hypothalamus, limbic system, subcortical and spinal motor areas were determined.

Up to now, no study has investigated the prevalence of vitamin d deficiency in patient with Alzheimer's disease. Our aim is to investigate the prevalence of vitamin D deficiency and analysis the associated characteristics in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have Alzheimer's dementia and their diagnosis must be made according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer Disease and Related Disorders Association (NINCDS/ADRDA) and DSM-IV criteria
* The informed consent form must be given by patients and/or their representatives

Exclusion Criteria:

* if the causes of dementia (lewy body dementia, vascular dementia, pick disease, frontotemporal dementia...) is out of Alzheimer's dementia,
* having chronic liver disease and/or end-stage renal disease
* if the informed consent form is being withdrawn

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with Alzheimer's dementia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D levels | January, 1, 2013

CONTACTS AND LOCATIONS:
Overall Officials: Ilkin M Naharci, specialist, Study Director — Gulhane Medical Faculty Training Hospital, Department of Internal Medicine, Division of Geriatrics
Locations (1):
- Gulhane Medical School Training Hospital, Ankara, Turkey (Türkiye)